CLINICAL TRIAL: NCT01215916
Title: A Phase 1b Study of LY573636-sodium in Combination With Alimta (Pemetrexed) in Patients With Solid Tumors
Brief Title: A Phase 1 Study in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11158; H8K-MC-JZAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors
Keywords: Solid tumors
MeSH Terms: interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: Pemetrexed followed by LY573636 (Experimental): Pemetrexed on Day 1 followed by LY573636 on Day 4
  Interventions: Drug: LY573636; Drug: Pemetrexed
- Experimental: LY573636 followed by Pemetrexed (Experimental): LY573636 on Day 1, pemetrexed on Day 4
  Interventions: Drug: LY573636; Drug: Pemetrexed
- Experimental: LY573636 and Pemetrexed on Day 1 (Experimental): LY573636 and Pemetrexed on Day 1
  Interventions: Drug: LY573636; Drug: Pemetrexed

INTERVENTIONS:
Drug: LY573636 — Individualized dose is dependent on a patient's height, weight, and gender and is adjusted to target a specific exposure range corrected for a patient's laboratory parameters. Intravenous dosing is completed once per cycle (cycle equals either 21 or 28 days).
  Patients may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Patients are pretreated with folic acid [350 micrograms (µg) to 1000 µg orally, daily], Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone [4 milligrams (mg) orally, twice daily or equivalent].
  Other Names: Tasisulam
Drug: Pemetrexed — 375 to 500 milligrams per square meter (mg/m^2), intravenous dosing is completed once per cycle (cycle equals either 21 or 28 days).
  Patients may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Patients are pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent).
  Other Names: LY231514; Alimta

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) regimen for the combination therapy of LY573636 and pemetrexed that may be safely administered to patients with a solid tumor that is not amenable to curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* You must have a diagnosis of a solid tumor malignancy that is not amenable to curative therapy
* You must have a serum albumin level greater than or equal to 3.0 grams per deciliter (g/dL) [30 grams per liter (g/L)]
* You must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* You must be reliable and willing to make yourself available for the duration of the study and are willing to follow study procedures
* Patients with reproductive potential should use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drugs
* Your test results assessing the function of your blood, kidneys, liver, and heart are satisfactory
* You must be willing to take folic acid, Vitamin B12, or prophylactic steroids
* You must able to interrupt the use of aspirin (other than an aspirin dose less than or equal to 1.3 grams per day) and/or other nonsteroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents, such as piroxicam)
* You must have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, hormone therapy, or other investigational therapy for at least 4 weeks (6 weeks for mitomycin-C or nitrosoureas) before study enrollment and recovered from the acute effects of therapy (except alopecia). Patients who have received whole-brain radiation must wait 90 days before starting study therapy.
* You must sign an informed consent

Exclusion Criteria:

* You cannot have received other investigational drugs within the last 30 days
* You cannot have other on-going serious illnesses including active bacterial, fugal, or viral infections
* You cannot require regular, periodic paracentesis or thoracentesis
* You cannot have active brain metastasis
* You cannot currently be receiving warfarin (Coumadin®) therapy
* You cannot be pregnant or lactating
* You cannot have received prior pemetrexed or LY573636
* You cannot have a second primary malignancy that could affect interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon.-Fri. 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study planned for dose-escalation followed by dose-confirmation phase. Enrollment stopped before anyone entered dose-confirmation phase. Participant (pt) Flow presents pt disposition during dose-escalation & provide reasons for pts who discontinued treatment. All pts who received atleast 1dose of study drug were considered to have completed study.
Groups:
- LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day 1: Participants received a combination of LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 300 µg/mL and 375 mg/m2 of pemetrexed administered IV over 10 minutes both on Day 1 of a 21-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1: Participants received a combination of LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 340 µg/mL and 500 mg/m2 of pemetrexed administered IV over 10 minutes both on Day 1 of a 21-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4; LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4: Participants received a combination of LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 300 µg/mL on day 1 and 375 mg/m2 of pemetrexed administered IV over 10 minutes on Day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4: Participants received a combination of LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 320 µg/mL on day 1 and 500 mg/m2 of pemetrexed administered IV over 10 minutes on Day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4: Participants received a combination of 375 mg/m2 of pemetrexed administered IV over 10 minutes on Day 1 and LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 300 µg/mL on day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4: Participants received a combination of 375 mg/m2 of pemetrexed administered IV over 10 minutes on Day 1 and LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 320 µg/mL on day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4: Participants received a combination of 500 mg/m2 of pemetrexed administered IV over 10 minutes on Day 1 and LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 320 µg/mL on day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
- Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4: Participants received a combination of 375 mg/m2 of pemetrexed administered IV over 10 minutes on Day 1 and LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 340 µg/mL on day 4 of a 28-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
Period: Overall Study
Arm/Group | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day 1 | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4
Started | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2
Received at Least 1 Dose of Either Drug | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2
Not completed — Progressive Disease | 0 | 2 | 1 | 2 | 5 | 4 | 5 | 3 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants: those who received 1 or more doses of LY573636 or pemetrexed.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day 1 | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4 | Total
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.63 (NA) — Only one participant was involved in this group, the SD is not applicable | 63.13 (11.54) | 60.36 (9.39) | 60.91 (10.47) | 59.52 (11.00) | 58.26 (6.22) | 50.50 (14.55) | 65.26 (5.80) | 68.27 (0.07) | 59.02 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 4 | 4 | 4 | 5 | 2 | 0 | 26
  Male | 0 | 0 | 2 | 2 | 2 | 0 | 4 | 1 | 2 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 4
  Caucasian | 1 | 5 | 3 | 5 | 6 | 3 | 7 | 2 | 2 | 34
  East Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2 | 39

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose
Description: Based on maximum tolerated dose (MTD) in Cycle 1: highest dose where <33% participants (pts) had dose-limiting toxicity (DLT). DLTs were adverse events (AE) possibly related to study drug or AEs that met any of National Cancer Institute's (NCI) Common Terminology Criteria for AEs (CTAE): Grade (G) 4 neutropenia lasting ≥5 days; G4 neutropenia with fever, G4 thrombocytopenia, G3 thrombocytopenia with bleeding, ≥G3 non-hematologic toxicity (except nausea/vomiting and diarrhea controlled by medication; electrolyte toxicity resolved with standard replacement treatment; alopecia; and elevated alanine aminotransferase or aspartate aminotransferase with preexisting hepatic metastasis, if agreed by investigator). Investigators, with sponsor, could declare a DLT if pt experienced increasing toxicity during treatment and it was clear that further treatment would expose pt to excessive risk. Enrollment was stopped during the dose-escalation phase, thus further dose-escalation was not explored.
Time Frame: Baseline to toxicity [up to end of Cycle 1 (cycle = 21 or 28 days)]
Population: Enrollment was stopped during the dose-escalation phase and it was too early to assess the recommended dose for Phase 2 or to estimate the MTD, therefore zero participants were analyzed.
Groups:
- Pemetrexed Followed by LY573636: Pemetrexed on Day 1 and LY573636 on Day 4.
  LY573636: Individualized dosing was dependent on a participant's height, weight, and gender and was adjusted to target a specific LY573636 concentration corrected for a participant's laboratory parameters. The targeted drug concentration range for LY573636 dosing was 300 micrograms per milliliter (ug/mL) up to 360 µg/mL. Intravenous dosing was completed once each 28-day cycle.
  Pemetrexed: 375 milligrams per square meter (mg/m^2) to 500 mg/m^2; intravenous dosing was completed once each 28-day cycle.
  Participants were pretreated with folic acid [350 micrograms (µg) to 1000 µg orally, daily], Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone [4 milligrams (mg) orally, twice daily or equivalent].
  Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- LY573636 Followed by Pemetrexed: LY573636 on Day 1 and pemetrexed on Day 4.
  LY573636: Individualized dosing was dependent on a participant's height, weight, and gender and was adjusted to target a specific LY573636 concentration corrected for a participant's laboratory parameters. The targeted drug concentration range for LY573636 dosing was 300 ug/mL up to 360 µg/mL. Intravenous dosing was completed once each 28-day cycle.
  Pemetrexed: 375 mg/m^2 to 500 mg/m^2; intravenous dosing was completed once each 28-day cycle.
  Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent).
  Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- LY573636 and Pemetrexed on Day 1: LY573636 and pemetrexed on Day 1.
  LY573636: Individualized dosing was dependent on a participant's height, weight, and gender and was adjusted to target a specific LY573636 concentration corrected for a participant's laboratory parameters. The targeted drug concentration range for LY573636 dosing was 300 ug/mL up to 360 µg/mL. Intravenous dosing was completed once each 21-day cycle.
  Pemetrexed: 375 mg/m^2 to 500 mg/m^2. Intravenous dosing was completed once each 21-day cycle.
  Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent).
  Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Arm/Group | Pemetrexed Followed by LY573636 | LY573636 Followed by Pemetrexed | LY573636 and Pemetrexed on Day 1
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects were defined as serious and other non-serious adverse events (AEs) regardless of causality. A summary of serious and all other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: Baseline to end of study (up to 1 year of treatment plus 30-day follow-up)
Population: All enrolled participants: those who received 1 or more doses of LY573636 or pemetrexed.
Measure: Count of Participants; unit: Participants
Arm/Group | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day 1 | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4
Number analyzed (Participants) | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2
Participants
  Serious AEs | 1 | 4 | 2 | 4 | 3 | 3 | 4 | 3 | 2
  Non-Serious AEs | 1 | 5 | 3 | 6 | 6 | 4 | 9 | 3 | 2

3. Secondary Outcome: Percentage of Participants With a Tumor Response
Description: Tumor response was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria and confirmed by repeat assessment. Complete Response (CR) was defined as the disappearance of all target lesions and the normalization of tumor marker levels for non-target lesions; Partial Response (PR) was defined as at least a 30% decrease in the sum of the longest diameter of target lesions. Percentage of participants with a tumor response = (number of participants with CR or PR/number of enrolled participants)*100.
Time Frame: Baseline to progressive disease (up to 1 year of treatment plus 30-day follow-up)
Population: All enrolled participants: those who received 1 or more doses of LY573636 or pemetrexed.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed Followed by LY573636 | LY573636 Followed by Pemetrexed | LY573636 and Pemetrexed on Day 1
Number analyzed (Participants) | 18 | 15 | 6
percentage of participants | 0.0 | 13.3 | 0.0

4. Secondary Outcome: Pharmacokinetics, Concentration Maximum (Cmax) of LY573636
Time Frame: Cycles 1 and 2 on Day 4 (prior to and at the end of LY573636 infusion, 2 and 4 hours post LY573636 infusion), Day 8 (anytime), Day 15 (anytime)
Population: Participants who had at least 1 evaluable Cmax pharmacokinetic sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- All Enrolled Participants: Participants who received 1 or more doses of LY573636.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 37
micrograms per milliliter (µg/mL)
  Cycle 1 | 264.285 (18.465)
  Cycle 2: number analyzed (Participants) | 27
  Cycle 2 | 225.588 (24.061)

5. Secondary Outcome: Pharmacokinetics, Area Under the Curve (AUC) of LY573636
Description: Area under the concentration-time curve above the albumin corrected threshold (AUCalb) is provided for LY573636, which has been found to be highly bound to albumin. AUCalb is a surrogate measure of exposure to unbound (free) LY573636.
Time Frame: as for outcome 4
Population: Participants who had at least 1 evaluable AUCalb pharmacokinetic sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter (h*µg/mL)
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 36
hour*micrograms per milliliter (h*µg/mL)
  Cycle 1 | 132.783 (265.75)
  Cycle 2: number analyzed (Participants) | 23
  Cycle 2 | 68.813 (1840.9)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 1 year of treatment plus 30-day follow-up)
Description: Deaths due to progressive disease were not considered serious adverse events and are provided in the Participant Flow.
Groups:
- LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day1: Participants received a combination of LY573636 administered over a 2-hour intravenous (IV) infusion to target a Cmax of 300 µg/mL and 375 mg/m2 of pemetrexed administered IV over 10 minutes both on Day 1 of a 21-day cycle. Participants were pretreated with folic acid (350 µg to 1000 µg orally, daily), Vitamin B12 (1000 µg intramuscular injection every 9 weeks), and dexamethasone (4 mg orally, twice daily or equivalent). Participants continued on study drug (LY573636 and pemetrexed) until disease progression, unacceptable toxicity, or if any other withdrawal criteria were met.
Arm/Group | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day1 | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4
Serious Adverse Events (participants affected / at risk) | 1/1 | 4/5 | 2/3 | 4/6 | 3/6 | 3/4 | 4/9 | 3/3 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 5/5 | 3/3 | 6/6 | 6/6 | 4/4 | 9/9 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day1 (N=1) | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 (N=5) | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 (N=3) | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 (N=6) | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 (N=6) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 (N=4) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 (N=9) | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 (N=3) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4 (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY573636, 300µg/mL Plus Pemetrexed, 375mg/m2 on Day1 (N=1) | LY573636, 340 µg/mL Plus Pemetrexed, 500 mg/m2 on Day 1 (N=5) | LY573636, 300 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 (N=3) | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 375 mg/m2 on Day4 (N=6) | LY573636, 320 µg/mL on Day1 Plus Pemetrexed, 500 mg/m2 on Day4 (N=6) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 300 µg/mL on Day4 (N=4) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 (N=9) | Pemetrexed, 500 mg/m2 on Day1 Plus LY573636, 320 µg/mL on Day4 (N=3) | Pemetrexed, 375 mg/m2 on Day1 Plus LY573636, 340 µg/mL on Day4 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (5) | 2 (5) | 2 (10) | 0 (0) | 3 (9) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (5) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (9) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (5) | 0 (0) | 2 (6) | 2 (4) | 0 (0) | 2 (3) | 1 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (5) | 3 (3) | 3 (9) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 3 (4) | 2 (4) | 2 (4) | 1 (5) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (5) | 3 (3) | 1 (3) | 1 (3) | 2 (4) | 5 (7) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periproctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (11) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 4 (11) | 2 (11) | 4 (11) | 3 (8) | 2 (4) | 5 (11) | 1 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (7) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 1 (2) | 1 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Spinal pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0/1 (0) | 0/4 (0) | 1/4 (1) | 0 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (10) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (8) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (9) | 1 (3) | 2 (5) | 0 (0) | 1 (3)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine colour abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (10) | 3 (6) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 2 (2) | 1 (6) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (13) | 2 (5) | 2 (6) | 0 (0) | 3 (5) | 2 (5) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (4) | 3 (7) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (2) | 1 (3) | 2 (4) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 2 (6) | 0 (0) | 2 (7) | 1 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (5) | 2 (2) | 0 (0) | 4 (8) | 1 (2) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (3) | 1 (4) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (7) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/1 (3) | 0/4 (0) | 0/4 (0) | 0 (0) | 1/5 (4) | 0/2 (0) | 0/0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0/1 (0) | 0/4 (0) | 0/4 (0) | 0 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0/1 (0) | 0/4 (0) | 0/4 (0) | 0 (0) | 0/5 (0) | 0/2 (0) | 0/0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (8) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (6) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrostomy tube placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was stopped early during dose-escalation phase. Original protocol dosed LY573636 and pemetrexed on Day 1; 21-day cycle. Protocol amended (due to dose limiting toxicities); LY573636 and pemetrexed doses separated by 3 days; 28-day cycle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days